CLINICAL TRIAL: NCT07116915
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics for a Single Dose of HRS-9821 Aerosol Inhaler Administered in Healthy Subjects and Multiple Doses in Patients With COPD
Brief Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics for a Single Dose of HRS-9821 Powder for Inhalation Administered in Healthy Subjects and Multiple Doses in Patients With COPD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-9821-I-102
Record Dates: First submitted 2025-07-22; First posted 2025-08-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HRS-9821 Powder for Inhalation (Experimental): Participants inhaled HRS-9821 powder either as a single dose or for 12 days.
  Interventions: Drug: HRS-9821 Powder for Inhalation.
- HRS-9821 Powder for Inhalation placebo (Placebo Comparator): Participants received a single dose or 12 consecutive days of inhaled powdered placebo with HRS-9821.
  Interventions: Drug: HRS-9821 Powder for Inhalation placebo
- Moxifloxacin (Active Comparator): Moxifloxacin is oral
  Interventions: Drug: Moxifloxacin Hydrochloride Tablets

INTERVENTIONS:
Drug: HRS-9821 Powder for Inhalation. — HRS-9821 Powder for Inhalation.
  Arms: HRS-9821 Powder for Inhalation
Drug: HRS-9821 Powder for Inhalation placebo — HRS-9821 Powder for Inhalation placebo
  Arms: HRS-9821 Powder for Inhalation placebo
Drug: Moxifloxacin Hydrochloride Tablets — Moxifloxacin Hydrochloride Tablets
  Arms: Moxifloxacin

SUMMARY:
The aim of this study was to evaluate the safety and tolerability of HRS-9821 Powder for Inhalationadministered in a single dose in healthy individuals and multiple doses in patients with COPD。

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was obtained to participate in the trial
2. Body weight ≥45 kg, BMI 18-33 kg/m2 (both ends included)
3. The 12-lead ECG was normal or abnormal but clinically insignificant until randomization
4. Contraception was strict from the time informed consent was signed until 1 month (for subjects receiving HRS-9821/ placebo) or 3 months (for male subjects receiving moxifloxacin) after the last dose
5. All study regulations and procedures were followed and inhalation devices used in the study were used correctly during the study

   The following inclusion criteria apply only to healthy subjects:
6. Vital signs were normal at screening
7. Pulmonary function was normal during screening
8. No smoking or smoking cessation ≥12 months before screening, and previous smoking history <5 pack-years；
9. Healthy male 18-50 years old The following inclusion criteria apply only to subjects with COPD
10. Male or female, aged 40-75 years;
11. Patients diagnosed with COPD;
12. A post-bronchodilator FEV1 /FVC < 0.7,40% ≤FEV1 < 80% of the predicted value,;
13. Smoking history of≥ 10 pack-years;
14. Normal chest X-ray examination results at screening;
15. Supporting discontinuation of COPD-related medications before randomization；

Exclusion Criteria:

1. Mean QTcF ≥ 450 ms at screening；
2. Persons who had donated blood or had massive blood loss (> 400 ml) within 4 weeks before screening or who were interested in donating blood during the study
3. Receipt of the investigational drug or device within 4 weeks before randomization or less than 5 times the half-life of the drug, whichever was greater;
4. Patients who had difficulty in blood collection or could not tolerate venipuncture in the past, such as dizzy with needles or blood
5. History of malignancy in any organ system
6. Known allergies to salbutamol, study medication, or any excipients in the formulation
7. Known previous infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); Or positive HIV (according to a trial-site SOP), treponema pallidum antibody, HBV surface antigen, or HCV antibody before randomization
8. History of alcohol abuse
9. History of drug abuse and drug dependence in the past 5 years；
10. Positive for alcohol or substance abuse test before randomization
11. During the study, surgery or treatment that might interfere with the conduct of the study was planned；
12. Unable or unwilling to fully adhere to the study protocol
13. Mentally or legally incapacitated
14. There were any other reasons for the subject not to participate in the study in the opinion of the investigator;
15. Use of a strong/moderate potency drug that inhibits or induces the hepatic drug-metabolizing enzyme CYP3A4 14 days before the first dose;
16. Drugs with effects on P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) were anticipated to be used during the study;
17. History of using HRS-9821 suspension;

    The following exclusion criteria apply only to healthy subjects:
18. Have been treated with antibiotics for upper and lower respiratory tract infections within 12 weeks prior to screening;
19. Abnormal laboratory or physical examination results with clinical significance;
20. Positive urine nicotine test before randomization;
21. Have consumed a prescription within 14 days prior to the first dose or over-the-counter drugs within 48 h prior to the first dose; The following exclusion criteria apply only to subjects with COPD
22. History of life-threatening acute exacerbation of COPD (AECOPD), including admission to intensive care unit and/or need for invasive ventilator support;
23. Diagnosed with other respiratory disorders;
24. Pulmonary heart disease, or pulmonary hypertension caused by lung disease and/or hypoxia;
25. History of lung volume reduction surgery, partial lung resection, lung transplantation, and other surgeries that may affect pulmonary function results;
26. History of AECOPD requiring systemic glucocorticoids or antibiotics or hospitalization within 4 weeks prior to screening;
27. Lower respiratory tract infection requiring antibiotic treatment within 4 weeks prior to screening;
28. Requiring oxygen therapy or home non-invasive ventilation;
29. Currently using or plan to use non-selective beta blockers or other drugs with bronchoconstrictive effects during the study;
30. Patients with serious trauma or major surgery within 6 months prior to screening who are still in the recovery period;
31. Abnormal laboratory tests at screening and baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the rate of adverse events | The screening period lasted until 40 days after administration

SECONDARY OUTCOMES:
Plasma drug concentration after administration | The screening period lasted until 40 days after administration
Changes in heart rate from baseline after a single dose of HRS-9821 aerosol inhalation in healthy subjects。 | The screening period lasted until 29 days after administration
Changes in QT interval from baseline after a single dose of HRS-9821 aerosol inhalation in healthy subjects. | The screening period lasted until 29 days after administration
Lung epithelial lining fluid (ELF) drug concentrations based on alveolar lavage (BAL) measurements in healthy subjects after a single dose of HRS-9821 aerosol inhalation | The screening period lasted until 29 days after administration
Theoretical intracellular drug concentrations based on alveolar lavage fluid (BALF) cells measured by alveolar lavage (BAL) after a single dose of HRS-9821 aerosol inhalation in healthy subjects. | The screening period lasted until 29 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided